CLINICAL TRIAL: NCT03122470
Title: Assessment of Advanced Imaging Techniques in the Evaluation and Management of Prostate Cancer
Brief Title: Correlation of Imaging Findings With Clinical Findings and Patient Outcomes in Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI departure - study not conducted.
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE10815
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
Keywords: TRUS biopsy; Pelvic MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MRI guided biopsy + TRUS biopsy (Experimental): Patients will undergo an MRI guided biopsy and standard trans-rectal ultrasonography-guided (TRUS) biopsy. Results will be compared to see which can more accurately diagnose and manage prostate cancer
  Interventions: Device: MRI guided biopsy; Procedure: TRUS biopsy

INTERVENTIONS:
Device: MRI guided biopsy — The MRI guided biopsy will preferentially be performed using a 3 tesla (3T) Siemens Verio, or 3T Siemens Skyra machine. The multiparametric MRI exam will consist of T1-, T2- and diffusion weighted imaging with or without post-contrast perfusion studies. magnetic resonance fingerprinting (MRF) will be performed before contrast injection. The MRI will be interpreted by two specified radiologists from the research team.
  Other Names: Prostate MRI; Pelvic MRI
Procedure: TRUS biopsy — The TRUS biopsy will be performed per current standard of care. Biopsy cores will be sent to pathology in separately labeled specimen cups. The final pathological results will be compared with pre-biopsy MRI findings.
  Other Names: Prostate Biopsy

SUMMARY:
MRI is being increasingly relied upon for detection, staging and management of prostate cancer. In this study patients with risk of prostate cancer will be recommended to have a pelvic MRI prior to the standard biopsy of the prostate and standard treatment of any detected prostate cancer. The results of the MRI will be compared to standard diagnosis techniques to see if cancer can be more accurately detected.

DETAILED DESCRIPTION:
The study team hypothesizes that strategic use of advanced MRI methods will provide a more accurate and less invasive approach for diagnosis and management of prostate cancer. The primary objectives are:

1. To develop advanced MRI methods and optimal MRI protocols for detection, staging, and follow-up of prostate cancer.
2. To evaluate the diagnostic performance of MRI-guided biopsy methods and correlate MRI findings with the pathological grade of cancer.
3. To correlate prostate MRI findings and biopsy results with patient progress and outcomes.
4. To evaluate the diagnostic accuracy of MRI in disease re-classification in patients on active surveillance.

Secondary Objectives:

1. To apply computer-aided advanced image analytic techniques (Computer-assisted diagnostics- CAD) to extract MRI features of patient clinical scans that correlate with diagnosis and grade of prostate cancer.
2. To study MRI features of lesions that mimic prostate cancer on imaging eg - chronic prostatitis, post treatment changes.
3. To evaluate the impact of MRI in decision making and choice of treatment by physicians and patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a suspicion (elevated PSA and/or abnormal digital rectal exam)/ diagnosis of prostate cancer

Inclusion criteria for sub-group follow-up scans:

1a. Patients who have undergone standard TRUS biopsy or TRUS with targeted biopsy (i.e cognitive TRUS, MR-TRUS fusion or TRUS + in-gantry biopsy)

Exclusion Criteria:

* Patients with ferromagnetic or otherwise non-MRI compatible aneurysm clips.
* The presence of an implanted pacemaker or implanted defibrillator device.
* Patients with contraindications for MRI due to embedded foreign metallic objects. Bullets, shrapnel, metalwork fragments, or other metallic material adds unnecessary risk to the patient.
* Implanted medical device not described above that is not MRI-compatible;
* Known history of severe claustrophobia;
* For patients with known history of allergic reaction to magnetic resonance (MR) contrast material or abnormal kidney function (glomerular filtration rate (GFR) < 30 mL/min), a contrast enhanced exam will not be performed; however, a non-contrast exam may be performed;
* Minors will be excluded.
* Prisoners and members of other vulnerable populations will be excluded from this study as these populations will not provide any additional unique information to or uniquely benefit from the study.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Number of patients with the most likely diagnosis based on the five-point scale - PIRADS | Up to two weeks after MRI
  Prostate imaging reporting and data system (PIRADS) scale: 1. Benign; 2. Probably benign; 3. Indeterminate; 4. Probably malignant; 5. Malignant
Number of patients with true diagnosis based on biopsy pathology | Up to two weeks after MRI
  1. Benign; 2. Probably benign; 3. Indeterminate; 4. Probably malignant; 5. Malignant

SECONDARY OUTCOMES:
biopsy and MRI based diagnosis match in at least 8/10 patients | Up to two weeks after MRI
  The score based on the true diagnosis and most likely diagnosis as agreed on by classifiers is the same in at least 80% of patients
Ratio of positive diagnosis as detected by pelvic MRI guided biopsy compared to standard TRUS biopsy | Up to two weeks after MRI
  The diagnostic performance of MRI guided biopsy techniques will be compared with standard TRUS biopsy using a single sample of patients undergoing both biopsy techniques. It has been reported that MRI consistently detects a larger number of clinically significant prostate cancers (sensitivity - 0.91 for MRI-guided biopsy vs 0.76 for TRUS biopsy), while avoiding the detection of cancers that are clinically insignificant, as compared to TRUS biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ponsky, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center